CLINICAL TRIAL: NCT03358082
Title: Effectivness of Topical Tacrolimus 0.03% Monotherapy in Patients With Vitiligo: Arandomized Controlled Trial
Brief Title: Effectivness of Topical Tacrolimus Monotherapy in Patients With Vitiligo
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aml Abd Elaziz Ahmed, Dermatology Resident in Farshot General Hospital, Qena, Egypt, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tacvit01
Record Dates: First submitted 2017-11-12; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Vitiligo; Tacrolimus
MeSH Terms: conditions — Vitiligo | interventions — Tacrolimus; Ointments; hydrocortisone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus group (Active Comparator): Tacrolimus 0.03% ointment twice daily for 6 months
  Interventions: Drug: Tacrolimus 0.03% Ointment
- Hydrocortisone group (Active Comparator): hydrocortisone acetate 1% ointment twice daily for 6 months
  Interventions: Drug: Hydrocortisone Acetate 1% Ointment

INTERVENTIONS:
Drug: Tacrolimus 0.03% Ointment — topical tacrolimus 0.03% twice daily for 6 months
  Other Names: Tarolimus ointment
  Arms: Tacrolimus group
Drug: Hydrocortisone Acetate 1% Ointment — hydrocortisone acetate 1% ointment twice daily for 6 months
  Other Names: Texacort ointment
  Arms: Hydrocortisone group

SUMMARY:
The study will evaluate the effectiveness of Tacrolimus 0.03% ointment monotherapy in patients with vitiligo. Patients will be treated for 6 months and followed for 3 months after treatment. All types of vitiligo will be included.

DETAILED DESCRIPTION:
Study approval: The study was submitted for approval by Scientific and Ethical Committee at Faculty of Medicine, Sohag University. An informed written consent will be obtained from all participants.

Study design: randomized controlled trial. Study population: the study will include patients who attend the outpatient Clinic of Dermatology & Venereology and Andrology, Faculty of Medicine, Sohag University in corporation with Farshot General Hospital. Women who are pregnant or lactating, children aged 2 years or less and patients with acute or chronic disease that might affect skin barrier function will be excluded.

Patients and methods:

Study participants will be randomly divided into two treatment groups: group A will receive 0.03% tacrolimus ointment and group B will receive hydrocortisone acetate 1% ointment twice daily for 6 months.

Patients will be evaluated at baseline and monthly intervals for 6 months and at 3 months after stopping treatment.

ELIGIBILITY:
Inclusion Criteria:

* all patients with clinical diagnosis of vitiligo

Exclusion Criteria:

* children =or <2 years old, women who are pregnant or lactating, patients with acute or chronic disease that might affect skin barrier function.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Vitiligo Area Scoring Index (VASI) | basline to 9 months
  * The percentage of vitiligo involvement for each body region is calculated by using the palmar method. The palmar method uses the palmar surface area of the patient's hand as an estimation guide and defines the surface of the patient's hand including fingers to be 1% of the total body surface area.
  * The extent of residual depigmentation is expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%.
  * At 100% depigmentation, no pigment is present; at 90%, specks of pigment are present; at 75%, the depigmented area exceeds the pigmented area; at 50%, the depigmented and pigmented areas are equal; at 25%, the pigmented area exceeds the depigmented area; at 10%, only specks of depigmentation are present.
  * VASI= ∑ [HAND UNITS] × [RESIDUAL DEPIGMENTATION].

SECONDARY OUTCOMES:
Vitiligo Disease Activity (VIDA) Score | baseline to 9 months
  ): is a six-point scale for evaluating vitiligo activity.
  * In this score grading is based on disease activity and time period. Grading is as follows: + 4: (activity lasting 6 weeks or less); score +3: (activity lasting 6 weeks to 3 months); score 2: (activity lasting 3-6 months); score1: (activity lasting 6-12 months); score 0: (stable for 1 year or more); score -1: (stable with spontaneous repigmentation for 1 year or more).
  * A low Vitiligo disease activity score indicate less vitiligo activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan Saleh, MD, Study Director — Sohag Faculty of Medicine, Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided